CLINICAL TRIAL: NCT07025278
Title: The Effects and Mechanisms of Game-based Cognitive-motor Dual-task Intervention on Fall Prevention Among Older Adults
Brief Title: The Effects of Cognitive-motor Dual-task Intervention on Fall Prevention Among Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jinyao Wang (Other)
Responsible Party: Sponsor-Investigator, Jinyao Wang, Principal Investigator, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Ethics No. 2573, 2024
Record Dates: First submitted 2025-06-01; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: ELDERLY PEOPLE; Cognitive-motor Dual-task; Fall Prevention; Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Medium difficulty fixed priority group (Experimental): Participants in this group underwent a medium-difficulty and fixed-priority cognitive-motor dual-task fall prevention intervention program
  Interventions: Behavioral: Medium difficulty fixed priority group
- Medium difficulty variable priority group (Active Comparator): Participants in this group underwent a medium-difficulty and variable-priority cognitive-motor dual-task fall prevention intervention program
  Interventions: Behavioral: Medium difficulty variable priority group

INTERVENTIONS:
Behavioral: Medium difficulty fixed priority group — During the intervention process, participants carried out cognitive and motor tasks simultaneously. They were told to divide attention equally between them and not prioritize one over the other.
  Arms: Medium difficulty fixed priority group
Behavioral: Medium difficulty variable priority group — During the intervention process, participants performed medium-difficulty cognitive and motor tasks simultaneously. Participants alter focus between the motor task and the cognitive task every half of the intervention time.
  Arms: Medium difficulty variable priority group

SUMMARY:
1. Develop an evidence-based dual-task intervention programme incorporating gamification for fall risk reduction in older adults.
2. Examine the effects of the gamified dual-task intervention on fall risk in older adults.
3. Elucidate the underlying mechanisms of the optimal gamified dual-task intervention programme in reducing falls in older adults.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old;
2. Able to walk independently for at least 10 meters without obvious pain or difficulty;
3. Free from lower limb and foot deformities, wounds, ulcers, or other diseases, and capable of wearing flexible devices;
4. Scored as low or moderate fall risk on the Morse Fall Risk Assessment Scale;
5. Scored > 40 points on the Berg Balance Scale and < 20 seconds on the Time Up and Go Test (TUG);
6. Scored ≥ 21 points on the Mini-Mental State Examination (MMSE);
7. With an educational level of primary school or above, able to correctly understand instructions and make corresponding responses;
8. Without diseases that severely affect cognitive and motor functions, including cardiovascular diseases (such as uncontrolled hypertension, heart failure, etc.), neurological diseases (such as Parkinson's disease, stroke, epilepsy, etc.), musculoskeletal diseases (such as severe arthritis, recent fractures, etc.), etc.;
9. Normal vision and hearing or corrected to normal, without affecting the understanding of instructions and participation in interventions;
10. Conscious and able to understand the test requirements;
11. Able to understand and sign the informed consent form voluntarily, and willing to cooperate in completing the research procedures.

Exclusion Criteria:

1. Must rely on assistive walking devices or others to walk;
2. Individuals with color vision disorders, including various types of color blindness and color weakness;
3. Unable to correctly perform addition and subtraction operations;
4. Those allergic to the materials of research equipment;
5. Currently participating in other research or intervention projects that may affect the effectiveness of this intervention.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
The changes of Time up and go test from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks

SECONDARY OUTCOMES:
The changes of the Berg Balance Scale (BBS) from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
  The minimum and maximum values of the Berg Balance Scale are 0 and 56 points, respectively. The higher the score, the better the balance ability, and the lower the risk of falling.
The changes of the Mini-Mental State Examination (MMSE) from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
  The minimum and maximum values of the Mini-Mental State Examination (MMSE) are 0 and 30 points, respectively. The higher the score, the better the cognitive function.
The changes of Trail making test from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
The changes of gait from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
  The gait of participants is measured using insole plantar pressure measurement systems to assess the step length, cadence, walking speed, and plantar pressure distribution. The results could determine whether gait abnormalities are present.

OTHER OUTCOMES:
The changes of the Falls Efficacy Scale-International (FES-I) from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
  The minimum and maximum values of the Falls Efficacy Scale-International (FES-I) are 16 and 64 points, respectively. A higher score indicates a greater degree of an individual's concern about falling.
The changes of 12-Item Health Survey from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
The changes of the Geriatric Depression Scale (GDS) from baseline to the end of the intervention | From enrollment to the end of the intervention at 3 weeks
  The minimum and maximum scores of the Geriatric Depression Scale (GDS) are 0 and 30 points, respectively. A higher score indicates more severe depressive symptoms in individuals.

IPD SHARING:
Plan to Share IPD: Undecided